CLINICAL TRIAL: NCT00130871
Title: Impact of Levosimendan Pretreatment on Weaning From Cardiopulmonary Bypass (CPB) in Patients With Diminished Left Ventricular Function Before Coronary Artery Bypass Grafting (CABG)
Brief Title: Levosimendan Pretreatment for Weaning Patients From Cardio-Pulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3001079; NCT00195832 (obsolete NCT alias)
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Heart Disease
Keywords: levosimendan; weaning; cardio-pulmonary bypass
MeSH Terms: conditions — Coronary Disease | interventions — Simendan

INTERVENTIONS:
Drug: levosimendan

SUMMARY:
The study evaluates the efficacy of intravenous levosimendan treatment started during a coronary artery bypass operation to wean patients from a heart lung machine.

DETAILED DESCRIPTION:
Levosimendan or placebo infusion is started at the time of induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Three vessel coronary artery disease.
* Indication for on-pump coronary artery bypass surgery.
* Ejection fraction below 50%

Exclusion Criteria:

* Indication for any cardiac valve surgery
* Previous coronary artery bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Proportion of successful primary weanings

CONTACTS AND LOCATIONS:
Overall Officials: Markku Salmenperä, MD, Principal Investigator — Helsinki University Central Hospital, Finland
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Central Hospital, Turku